CLINICAL TRIAL: NCT00727246
Title: CDP-Choline and Working Memory After TBI: A Neuroimaging Study.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Patricia M. Arenth (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Patricia M. Arenth, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PRO07020121; K23HD049626 (NIH)
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Results first posted 2017-07-28 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-06

CONDITIONS: Brain Injuries
Keywords: Traumatic Brain Injury; FMRI; Memory; Cognition; Neuropsychology
MeSH Terms: conditions — Brain Injuries; Brain Injuries, Traumatic | interventions — Cytidine Diphosphate Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CDP-Choline (Experimental): Treatment with CDP-Choline
  Interventions: Drug: CDP-Choline
- Placebo (Placebo Comparator): Treatment with Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDP-Choline — 1000 mg CDP-Choline 2 x per day for 6 weeks.
  Other Names: Citicoline; Cytidine 5'-diphosphocholine
  Arms: CDP-Choline
Drug: Placebo — Treatment with placebo for 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether an investigational drug, called "CDP-Choline", improves memory in people with traumatic brain injury (TBI). To do this, we are asking for people with traumatic brain injury and people without traumatic brain injury to be a part of this study. We will compare results between each group to see if this investigational drug makes a difference with memory. We will also compare brain imaging results and information collected before and after the taking of the study medication to see if there are any differences. We hypothesize that there will be differences in brain activation patterns between individuals with TBI and healthy controls, as well as differences in performance on memory testing at baseline. We further hypothesize that, after treatment with CDP-Choline, the patterns in neuroimaging findings and cognitive testing results for individuals with TBI will more closely resemble results observed for healthy individuals. We hope that what we learn from this study will be helpful in the future treatment of individuals with head injury.

DETAILED DESCRIPTION:
Despite the prevalence of working memory deficits following traumatic brain injury (TBI), the scientific data regarding pharmacological treatment of this problem is limited. As deficits in working memory are known to have a significant impact on functional outcomes for individuals with TBI, further research in this area is essential in order for physicians to be able to treat this problem more effectively. The primary goal of the proposed project is to examine the efficacy of a particular pharmacological agent, CDP-Choline, in the treatment of working memory deficits following traumatic brain injury (TBI). The study sample will consist of 48 subjects: A group of 24 individuals who have sustained moderate to severe TBI, and a group of 24 healthy controls. Each group will be divided into a placebo and treatment group. The project will utilize functional Magnetic Resonance Imaging (fMRI) to investigate the cerebral neurophysiological effects of treatment with CDP-Choline. A working memory task (N-Back) will be employed during fMRI sessions. In addition, the effects of treatment with CDP-Choline on neuropsychological testing performance will also be evaluated, and the correlations between behavioral performance and neuroimaging results will be observed. We will achieve these goals by comparing baseline neuropsychological testing results as well as fMRI results, with a second set of testing and neuroimaging results obtained following 1 month of pharmacological treatment with CDP Choline or placebo. Based on our preliminary studies and the available literature, we expect to see the following: Baseline fMRI results are expected to show that individuals with TBI display altered patterns of cerebral activation during a working memory task, as compared to healthy controls. With CDP-Choline treatment, we expect TBI subjects to display fMRI laterality and dispersion patterns that more closely resemble patterns of healthy controls. In addition, we anticipate improvements in behavioral performance on both the specific working memory task (N-Back), and on traditional neuropsychological tests to be associated with CDP-Choline treatment, with greater magnitude of change on testing results for the TBI group as compared to any changes noted for the control or placebo groups. Finally, we anticipate that specific significant correlations will be observed between neuropsychological testing results and neuroimaging findings, and that the strength of these relationships will be greater for the TBI treatment group, as compared to the placebo or healthy control groups. By conducting the proposed study in this manner, we hope to provide scientific data that will allow for improved treatment, and ultimately improved functional outcomes for individuals who have sustained TBI.

ELIGIBILITY:
Inclusion Criteria:

For individuals with TBI and Health Controls:

* right hand dominant
* English speaking
* No history of neurological illness (for example, stroke, seizure or brain tumor.
* No significant history of psychiatric illness (for example, schizophrenia or bipolar disorder) or current severe emotional distress.
* No visual difficulties that would not allow for reading and following written instructions.
* Free of alcohol or substance abuse.
* Capable of following basic written and oral instructions.
* Not taking certain medications that may interact with study medication or interfere with neuroimaging.
* Be able to take medication in tablet form, or crushed and dissolved in a liquid.
* Meet the additional criteria associated with MRI safety standards, as required by the University of Pittsburgh Department of Radiology. For example, these criteria include exclusion due to surgical placement of metal plates or electronic implants.

In addition:

Individuals with TBI must:

* Have a specific diagnosis of a moderate to severe traumatic brain injury, which can be confirmed through review of medical records or assessments.
* Be at least 1 year, but no more than 3 years since injury.
* Must have significant working memory problems, as indicated by performance on a screening test.

Normal Control subjects must:

* Perform within the normal range on a test of working memory.

Exclusion Criteria:

* Prisoners.
* Males with sexual partners who are planning to become pregnant during the treatment period.
* Females who are currently pregnant or who are planning to become pregnant during the treatment period.
* Individuals who are currently enrolled in another medication study
* Individuals who are currently, or have previously been, treated with CDP-Choline (Citicoline) for research or clinical purposes.
* Currently in a nursing home in the state of Pennsylvania.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2009-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patricia M. Arenth, Ph.D., Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Department of Physical Medicine & Rehabilitation, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Data collected was significantly limited

REFERENCES:
- See also: University of Pittsburgh School of Medicine, Department of Physical Medicine & Rehabilitation — http://www.rehabmedicine.pitt.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants With TBI Who Received CDP-Choline: Participants who have experienced a TBI and were randomly assigned to receive the study supplement
- Participants With TBI Who Received Placebo: Participants with a history of TBI who were randomly assigned to the placebo group
- Control Participants Who Received CDP-Choline: Individuals without a history of TBI who acted as control participants and were randomly assigned to receive CDP-Choline
- Control Participants Who Received Placebo: Individuals without a history of TBI who participated as control subjects and were randomly assigned to receive placebo
Period: Overall Study
Arm/Group | Participants With TBI Who Received CDP-Choline | Participants With TBI Who Received Placebo | Control Participants Who Received CDP-Choline | Control Participants Who Received Placebo
Started | 3 | 3 | 8 | 5
Completed | 3 | 2 | 7 | 3
Not Completed | 0 | 1 | 1 | 2
Not completed — could not complete MRI | 0 | 1 | 0 | 1
Not completed — incidental finding | 0 | 0 | 0 | 1
Not completed — withdrawn | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants With TBI Who Received CDP-Choline: Participants with TBI who were randomized to receive the CDP-Choline
- Participants With TBI Who Received Placebo: Participants with TBI who were randomized to receive Placebo
- Control Participants Who Received CDP-Choline: Participants without a history of TBI who were randomized to receive CDP-Choline
- Control Participants Who Received Placebo: Participants without a history of TBI who were randomized to receive placebo
- Total: Total of all reporting groups
Arm/Group | Participants With TBI Who Received CDP-Choline | Participants With TBI Who Received Placebo | Control Participants Who Received CDP-Choline | Control Participants Who Received Placebo | Total
Number analyzed (Participants) | 3 | 2 | 7 | 3 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.66 (12.42) | 25 (1.41) | 29 (7.90) | 34 (13) | 29.8 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 2 | 7
  Male | 2 | 1 | 4 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 3 | 2 | 7 | 3 | 15

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Composite Score for Group of Subjects With TBI and Healthy Controls Matched by Age, Education, and Treatment Group.
Description: .A mean index score created as a composite cognitive performance across domains. Purpose was to serve as a measure of overall cognitive functioning for data analysis. A higher T-score indicates a higher level of cognitive function. Due to matching criteria of age range, gender and education level, as well as the small number of subjects with TBI who complete the study (n = 5), matched groups required a reduction to 2 subjects per group for analysis as planned per protocol. Due to the small number of subjects in this study overall, although analyses were run, results should be considered with caution.
Time Frame: 6 weeks
Population: A repeated measure ANOVA was completed to evaluate potential differences in cognitive composite scores of subjects with TBI as compared to healthy controls 6 weeks after treatment with CDP Choline (1000 mg CDP-Choline 2 x per day for 6 weeks) as compared to those treated with placebo. Matching criteria and small n for TBI group reduced group sizes.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Participants With TBI Who Received CDP-Choline | Participants With TBI Who Received Placebo | Control Participants Who Received CDP-Choline | Control Participants Who Received Placebo
Number analyzed (Participants) | 2 | 2 | 2 | 2
T-score | 42.750 [27.163 to 58.337] | 50.500 [34.913 to 66.087] | 49.500 [33.913 to 65.987] | 55.000 [39.413 to 70.587]
Statistical Analysis 1: Comparison: Participants With TBI Who Received CDP-Choline vs Participants With TBI Who Received Placebo vs Control Participants Who Received CDP-Choline vs Control Participants Who Received Placebo; A repeated measures ANOVA was completed to evaluate differences in cognitive composite scores of individuals with a history of TBI as compared to healthy controls 6 weeks after treatment with CDP Choline (1000 mg CDP-Choline 2 x per day for 6 weeks) as compared to those treated with placebo. A mean index score created as a composite cognitive performance across domains (higher t-score = higher cognition). Purpose was to serve as a measure of overall cognitive functioning for data analysis; Test type: Other; p = .85, ANOVA; A repeated measures ANOVA was completed to evaluate differences in cognitive composite scores between groups and CDP-Choline or placebo

2. Primary Outcome: Cognitive Composite Score for Group of Subjects With TBI and Unmatched Healthy Controls
Description: A mean index score created as a composite cognitive performance across domains. Purpose was to serve as a measure of overall cognitive functioning for data analysis. Higher T-scores indicate higher levels of cognitive functioning. Due to the small number of subjects in this study, this second analysis was completed using the same number of subjects in the TBI and control groups, but without matching so that a slightly larger number of subject's data could be utilized. Although analyses were run, due to the very small number of participants in this study, results should be considered with caution.
Time Frame: 6 weeks
Population: cognitive composite scores of individuals with a history of TBI as compared to healthy controls 6 weeks after treatment with CDP Choline (1000 mg CDP-Choline 2 x per day for 6 weeks) as compared to those treated with placebo. See note above related to the limited number of subjects in each group.
Measure: Mean (95% Confidence Interval); unit: T-score
Arm/Group | Participants With TBI Who Received CDP-Choline | Participants With TBI Who Received Placebo | Control Participants Who Received CDP-Choline | Control Participants Who Received Placebo
Number analyzed (Participants) | 2 | 3 | 3 | 2
T-score | 55.750 [46.187 to 65.313] | 50.167 [42.358 to 57.975] | 53.000 [45.192 to 60.808] | 55.000 [45.437 to 64.563]
Statistical Analysis 1: Comparison: Participants With TBI Who Received CDP-Choline vs Participants With TBI Who Received Placebo vs Control Participants Who Received CDP-Choline vs Control Participants Who Received Placebo; A repeated measure ANOVA was completed to evaluate potential differences in cognitive composite scores of individuals with a history of TBI as compared to healthy controls 6 weeks after treatment with CDP Choline (1000 mg CDP-Choline 2 x per day for 6 weeks) as compared to those treated with placebo; Test type: Other; p = .329, ANOVA; [statistical method as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Participants With TBI Who Received CDP-Choline | Participants With TBI Who Received Placebo | Control Participants Who Received CDP-Choline | Control Participants Who Received Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 1/3 | 0/2 | 2/7 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants With TBI Who Received CDP-Choline (N=3) | Participants With TBI Who Received Placebo (N=2) | Control Participants Who Received CDP-Choline (N=7) | Control Participants Who Received Placebo (N=3)
Car Accident (Social circumstances) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headaches (daily) (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to multiple complex issues, recruitment was significantly lower than anticipated. As a result, statistical analyses are presented, however the number of subjects in each comparison group was very low and results should be considered with caution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes